CLINICAL TRIAL: NCT07071883
Title: Group Activities to Support Addiction Recovery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Nicholas Guenzel, Assistant professor, University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0449-24-FB
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Addiction; Substance Use Disorders (SUD)
Keywords: holotropic breathwork; addiction; recovery
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A--for individuals in residential treatment programs (Experimental): Arm A will use a cluster randomized intervention, providing HB for individuals at two facilities and a Multiple Modality (MM) intervention (yoga, meditation, and a film/discussion) at a third facility.
  Interventions: Behavioral: Holotropic breathwork; Behavioral: Multiple modality
- B--for individuals living in the community (Experimental): Arm B will be comprised of a single group and participants in this group will receive the same HB experience as the participants in the Arm A HB group
  Interventions: Behavioral: Holotropic breathwork

INTERVENTIONS:
Behavioral: Holotropic breathwork — HB is the practice of self-directed hyperventilation while lying down with the support of a selected music set and trained facilitators. Participants may experience an expanded state of consciousness with altered cognition, perception, and emotions.
Behavioral: Multiple modality — Multiple Modality (MM) intervention (yoga, meditation, and a film/discussion)
  Arms: A--for individuals in residential treatment programs

SUMMARY:
The purpose of this study is to pilot the use of Holotropic Breathwork (HB) for individuals seeking to recover from addiction. The study will have two arms: A--for individuals in residential treatment programs, B--for individuals living in the community. Arm A will use a cluster randomized intervention, providing HB for individuals at two facilities and a Multiple Modality (MM) intervention (soundbath, meditation, and a film/discussion) at a third facility. In Arm B, we seek to measure the feasibility, acceptability, and preliminary impact of HB among people with addiction living in the community. Arm B will be comprised of a single group and participants in this group will receive the same HB experience as the participants in the Arm A HB group. HB is the practice of self-directed hyperventilation while lying down with the support of a selected music set and trained facilitators. Participants may experience an expanded state of consciousness with altered cognition, perception, and emotions. HB has been associated improved mental functioning among the general public and people in addiction treatment, but has never been evaluated in a controlled trial. Inclusion criteria consist of being 19 years of age or older and having met criteria for a substance use disorder within the past five years. Additional inclusion criteria for participants in arm A include being in a residential addiction treatment program at CenterPointe or the Bridge.

Exclusion criteria form the Arm A HB group and the Arm B group include having been diagnosed with a bipolar disorder or a psychotic disorder or having had psychotic symptoms at any point in life, diagnosed with a cardiac condition, received care for a cardiac condition, or have current cardiac symptoms, ever diagnosed with a seizure disorder, current uncontrolled hypertension (140/90 or greater), diagnosed with glaucoma or retinal detachment, recent surgeries, or currently pregnant. Four breathwork sessions will be held: two at the UNMC College of Nursing in Lincoln, one at CenterPointe in Omaha, and one at The Bridge in Lincoln. One MM session will be held at The Bridge in Lincoln.

DETAILED DESCRIPTION:
This study evaluates the feasibility, safety, acceptability, and preliminary psychological and behavioral effects of Holotropic Breathwork (HB) as a supportive intervention for individuals in recovery from substance use disorders. HB is compared with a Multiple-Modality (MM) activity day in the residential setting. The study also assesses HB delivered to individuals in community-based recovery settings.

Study Overview

The project includes two primary participant groups:

Arm A - Residential Participants

Participants are recruited from two residential treatment programs (CenterPointe Omaha and The Bridge Lincoln). This arm uses cluster randomization: two sites will host the HB intervention, while an independent residential cohort at The Bridge will receive the MM intervention. Participants at each site receive the intervention assigned to their facility.

Arm B - Community Participants

Community members in addiction recovery are recruited via flyers, social media, and word-of-mouth. Arm B participants receive HB only and are included to evaluate feasibility, acceptability, and pre/post changes in functioning.

Across both arms, participants are evaluated at baseline, <24 hours post-intervention, and at 1-, 3-, and 6-month follow-up.

Rationale and Scientific Framework

Holotropic Breathwork is a structured, facilitator-led breathing practice designed to produce non-ordinary states of consciousness without the use of pharmacological agents. Prior research suggests HB may improve psychological, interpersonal, and existential functioning-domains strongly associated with addiction recovery.

Guided by conceptual models from psychedelic-assisted therapy research, this study hypothesizes that HB may elicit:

Mystical-type experiences

Challenging experiences

Emotional breakthroughs

These experiences may lead to psychological insight, which may contribute to improvements in mood, interpersonal relationships, existential wellbeing, and ultimately reductions in cravings or lapses.

Interventions Holotropic Breathwork (HB)

HB sessions may include up to 30 participants and follow a standardized protocol conducted by certified facilitators and trained apprentices (approximate facilitator-to-breather ratio 1:5).

HB events comprise the following elements:

Pre-Session Screening

Urine pregnancy test for participants who could become pregnant

Seated blood pressure measurement (must be <140/90)

Review of PHQ-9 to identify acute suicide risk

Assessment of medical and psychiatric exclusion criteria

Opening Circle

Participant introductions

Review of confidentiality, safety expectations, and session agreements

Educational Presentation (~60 minutes)

Content includes:

History and principles of HB

Hylotropic vs. holotropic states

Grof's cartography of the psyche (biographical, perinatal, and transpersonal domains)

COEX systems and emotional memory patterns

Strategies for navigating challenging experiences

Roles of breathers and sitters

Individual Readiness Check-ins Each participant meets briefly with a facilitator to assess emotional readiness and address questions.

Breathwork Session (~2 hours 20 minutes)

Participants lie on mats, typically using eyeshades

Guided relaxation prompts followed by intensified, self-paced breathing

Purposefully sequenced music supports the internal process

Sitters provide assistance only upon explicit request

Facilitators monitor safety continuously and may support participants through physical expressions of emotional release, ensuring all touch is participant-directed and consent-based

Post-Session Processing

Brief one-on-one check-ins with a facilitator

Participants may draw, write, or rest

Integration Presentation (~60 minutes)

Overview of formal and informal integration practices

Guidance on self-care, managing stimulation, and delaying major decisions

Discussion of appropriate sharing of HB experiences

Closing Circle Participants share reflections voluntarily; additional one-on-one support is available.

HB sessions conducted in Arm B follow the same structure and staffing.

Multiple-Modality (MM) Activity Day (Arm A Comparator)

The MM day is an attention-matched comparator condition designed to provide supportive, group-based activities without inducing non-ordinary states of consciousness. It is delivered only at The Bridge Lincoln.

The MM session includes:

Opening Circle Participants introduce themselves and may share recovery reflections.

Sound Bath Introduction Video (7 minutes) A brief educational video describing sound-based relaxation practices.

Sound Bath Session (20 minutes) Participants experience a guided sound bath in a quiet, low-stimulation environment.

Progressive Relaxation Exercise (11 minutes) A recorded body-relaxation sequence guides participants through calming techniques.

Film Screening (1 hour 43 minutes) Participants view Ben Is Back, a film depicting addiction and family dynamics.

Facilitated Group Discussion A trained UNMC nursing faculty member leads a structured conversation on themes from the film.

Closing Circle Participants may share insights or reflections before the session ends.

Unlike HB, MM activities pose no known physiological risks; therefore individuals excluded from HB remain eligible for the MM day.

Eligibility Criteria Inclusion Criteria

Adults aged 19 and older

Met criteria for a substance use disorder within the past 5 years

Arm A participants must be enrolled in residential treatment

Exclusion Criteria for HB (Arm A HB and Arm B)

Participants are excluded from HB if any of the following apply:

Lifetime diagnosis of bipolar disorder

Psychotic disorder or lifetime history of psychotic symptoms

Cardiac condition, history of cardiac treatment, or current cardiac symptoms

Seizure disorder

Uncontrolled hypertension (≥140/90)

Glaucoma or retinal detachment

Recent significant surgeries

Pregnancy

Acute suicidal ideation with plan or intent

These exclusions do not apply to MM participants.

Recruitment and Informed Consent Arm A (Residential)

The PI works with clinical staff to identify eligible residents. The PI delivers a standardized presentation, answers questions, and obtains individual informed consent in a private setting.

Arm B (Community)

Recruitment materials are posted through treatment centers, recovery organizations, and social media. Interested individuals contact the PI, receive study information, and complete consent via Zoom or in private at a participating site.

Data Collection and Outcome Measures

Assessments occur at:

Baseline

<24 hours post-session

1 month

3 months

6 months

Measures include:

Substance use: Timeline Followback, craving scale

Mental health: PHQ-9, GAD-7

Interpersonal functioning: SIFS

Existential functioning: PIL-SF

Psychological insight: PILS-6

Experiential measures: Mystical Experience Questionnaire, Challenging Experience Questionnaire, Emotional Breakthrough Inventory

Acceptability surveys

All follow-up surveys are administered through REDCap.

Safety Monitoring

Participant safety is supported by:

Continuous facilitator monitoring during HB sessions

Immediate exclusion of participants with elevated BP or positive pregnancy test

Real-time review of PHQ-9 scores by the PI

Same-day and next-day follow-ups for participants experiencing significant emotional reactions

Transportation assistance for participants who are physically unsteady

Emergency protocols including activation of emergency medical services when indicated

Stopping Rule

The study will be halted if more than 15% of participants require outside medical or psychiatric treatment related to the intervention.

Integration Support

HB participants are invited to attend two optional Zoom-based integration groups held:

5-7 days post-session

12-14 days post-session

Sessions are led by certified facilitators and apprentices. These groups offer guidance and reflection but do not involve data collection.

Statistical Analysis

Paired-samples t-tests will evaluate pre-post changes within HB participants.

Chi-square tests will compare cravings and lapses between HB and MM groups in Arm A.

Feasibility and acceptability metrics will include recruitment yield, attrition, survey completeness, and qualitative acceptability responses.

The study is not powered for definitive clinical outcomes but will provide effect-size estimates and procedural feasibility data to inform larger trials.

Potential Benefits and Risks

Participants may experience reductions in stress or anxiety, emotional release, heightened psychological insight, and enhanced purpose or meaning in life. Risks include temporary dizziness, emotional discomfort, recollection of traumatic events, and other transient psychological reactions. HB has a long history of safe use when conducted by certified facilitators.

ELIGIBILITY:
Inclusion Criteria:

* Arm A 19 years of age or older Currently enrolled in a residential addiction treatment program at CenterPointe or the Bridge Met criteria for a substance use disorder in the past five years
* Arm B 19 years of age or older Met criteria for a substance use disorder in the past five years

Exclusion Criteria:

* Arm A: HB group and Arm B

  1. Diagnosed with a bipolar disorder at any point in life (per self-report)
  2. Diagnosed with a psychotic disorder or have had psychotic symptoms at any point in life (per self-report)
  3. Diagnosed with a cardiac condition, received care for a cardiac condition, or have current cardiac symptoms (per self-report)
  4. Ever diagnosed with a seizure disorder (per self-report)
  5. Current uncontrolled hypertension (140/90 or greater) (measured the morning of the breathwork)
  6. Ever diagnosed with glaucoma or retinal detachment
  7. Recent surgeries
  8. Currently pregnant (individuals who have engaged in sexual activity since their last menstrual period will be asked to submit a urine sample for a pregnancy screen the morning of the breathwork)
  9. Acutely suicidal (i.e. with an intention and a plan)
* Arm A: MM group None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting a change in their substance use | 1 month, 3 months, and 6 months
  Timeline Followback (TLFB)

SECONDARY OUTCOMES:
Change in Psychological Insight | Baseline, <24 hours post-session, 1 month, 3 months, and 6 months
  Psychological Insight Scale (PILS-6)
Change in Depression Symptoms | Baseline, 1 month, 3 months, and 6 months
  Patient Health Questionnaire-9 (PHQ-9)
Change in Anxiety Symptoms | Baseline, 1 month, 3 months, and 6 months
  Generalized Anxiety Disorder-7 (GAD-7)
Change in Interpersonal Functioning | Baseline, 1 month, 3 months, and 6 months
  Self and Interpersonal Functioning Scale (SIFS)
Change in Purpose in Life | Baseline, 1 month, 3 months, and 6 months
  Purpose in Life Test - Short Form (PIL-SF)
Change in Cravings | Baseline, 1 month, 3 months, and 6 months
  Brief Craving Scale
Mystical Experiences | <24 hours post-session
  Mystical Experiences Questionnaire (MEQ)
Challenging Experiences | <24 hours post-session
  Challenging Experiences Questionnaire (CEQ)
Emotional Breakthrough | <24 hours post-session
  Emotional Breakthrough Inventory (EBI)
Acceptability of the Intervention | <24 hours post-session and 1 month
  Custom Acceptability Survey

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Arien Guenzel, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No